CLINICAL TRIAL: NCT04324138
Title: Efficacy and Safety of Jianpi Qinghua Granules in Patients With Nonerosive Reflux Disease:a Multicenter,Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Efficacy and Safety of Jianpi Qinghua Granules in Patients With Nonerosive Reflux Disease
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Liaoning University of Traditional Chinese Medicine (Other); First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019YFC1709602-
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Nonerosive Reflux Disease
Keywords: Nonerosive Reflux Disease; Traditional Chinese Medicine; Randomized placebo controlled trial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Jianpi Qinghua granules, 3 times a day and 1 hour after a meal
  Interventions: Drug: Jianpi Qinghua granules
- Control group (Sham Comparator): Jianpi Qinghua placebo granules(inclued 5% of experimental drug),3 times a day and 1 hour after a meal
  Interventions: Drug: Jianpi Qinghua placebo granules

INTERVENTIONS:
Drug: Jianpi Qinghua granules — 3 times a day and 1 hour after a meal, for 4 weeks
  Other Names: experimental drugs
  Arms: Experimental group
Drug: Jianpi Qinghua placebo granules — 3 times a day and 1 hour after a meal, for 4 weeks
  Other Names: placebo
  Arms: Control group

SUMMARY:
Nonerosive reflux disease (NERD) is a common refractory gastrointestinal disease. Proton pump inhibitors (PPIs), the first choice drug, have the following problems in clinical use: about 50 % of patients have no response to PPIs; the efficacy of simple acid suppression is poor; long-term use of PPIs can lead to indigestion, gastric polyps, atrophic gastritis, intestinal dysbacteriosis. Spleen Deficiency and Damp-heat Syndrome is one of the common clinical syndrome of NERD.TCM syndrome differentiation and treatment has the advantages of overall regulation and individualized treatment, but lack of high-level evidence. The purpose of this study is to evaluate the efficacy and safety of Jianpi Qinghua Granules for treating NERD with spleen deficiency and damp heat syndrome.

DETAILED DESCRIPTION:
Nonerosive reflux disease (NERD), representing about 70% of gastroesophageal reflux disease, is a common refractory gastrointestinal disease. Proton pump inhibitors (PPIs), the first choice drug, have the following problems in clinical use: about 50 % of patients have no response to PPIs; the efficacy of simple acid suppression is poor; long-term use of PPIs can lead to indigestion, gastric polyps, atrophic gastritis, intestinal dysbacteriosis. Spleen Deficiency and Damp-heat Syndrome is one of the common clinical syndrome of NERD.TCM syndrome differentiation and treatment has the advantages of overall regulation and individualized treatment, but lack of high-level evidence. NERD is the result of multifactorial pathogenicity. The reflux symptoms not only related to acid reflux, but also related to alkali, gas, mixed reflux, etc. The theory of Tongjiang put forward by Academician Dong Jianhua.Under the guidance of Academician Dong Jianhua, the research team create a prescription Jianpi Qinghua granule for treating NERD with spleen deficiency and damp-heat syndrome. The purpose of this study is to evaluate the efficacy and safety of Jianpi Qinghua Granules for treating NERD with spleen deficiency and damp heat syndrome based on a a multicenter,randomized, double-blind, placebo-controlled clinical trial.

On the basis of previous work, the project plans to establish sub centers in 3 Chinese hospitals, including78 patients with NERD and spleen deficiency and damp-heat syndrome. The therapeutic effects were evaluated from the following aspects: the VAS score of reflow and heartburn, the rate of discontinuation of antacids, the rate of recurrence of NERD symptoms, the score of TCM syndromes and the improvement of gastrointestinal function.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with non-erosive reflux disease
2. Subjects who have a medical history of PPI with poor therapeutic effect
3. Subjects aged between 18 and 70 years
4. Subjects diagnosed with spleen deficiency damp-heat syndrome of traditional Chinese medicine
5. Subjects who voluntarily signed written informed consent form

Exclusion Criteria:

1. Subjects who have active peptic ulcer, gastrointestinal hemorrhage, severe dysplasia of gastric mucosa or suspected malignant change, achalasia or postoperative achalasia
2. Subjects who have organic diseases of the digestive system (such as acute and chronic pancreatitis, cirrhosis, etc.), or systemic diseases that affect the gastrointestinal motility, such as hyperthyroidism, diabetes mellitus over 10 years, chronic renal insufficiency, spirit (the score of SAS and SDS shows severe anxiety or depression), nervous system diseases, etc
3. Subjects who have severe organ diseases such as heart, liver and kidney (such as ALT, AST more than 2 times of normal value), hematopoietic system diseases and tumors
4. Pregnant or lactating women
5. Subjects who have a history of nervous system disease and mental disease
6. Subjects who have a history of allergies to all the test drugs
7. Subjects who are participating in other clinical trials or have participated in other clinical trials within 4 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of visual analogue (VAS) score of reflux symptoms and heartburn | week 1, week 2，week 3, week 4 during treatment period, week 6 and week 8 during follow-up period
  During the treatment, the patients recorded the reflux and heartburn attacks (attack times and duration) within 24 hours every day on the symptom diary card, and VAS scores were performed on the reflux and heartburn symptoms. The average score of each symptom in the past week was calculated. The decrease rate of symptom score≥50% from baseline was recorded as response after 1 week of treatment , and the number of response weeks was more than 50% of the whole treatment period, which was considered effective.

SECONDARY OUTCOMES:
Change of secondary symptom score | week 2, week 4 during treatment period, week 6 and week 8 during follow-up period
  The secondary symptoms of Non-cardiogenic chest pain, epigastric pain, upper abdominal burning sensation, belching, cough, asthma, Pharyngeal different feeling were recorded. Each symptom was scored for frequency (score, 0-5) and severity (score, 0-5). A higher score represented more frequency and severity. Change of total symptom score from baseline was compared between treatment group and control group at different time windows . Reduction in total symptom score represented Improvement
Change of traditional Chinese Medicine syndrome score | week 2, week 4 during treatment period, week 6 and week 8 during follow-up period
  The symptoms related to spleen deficiency damp-heat syndrome were scored. The cardinal symptom was scored 0, 2, 4, 6 and the secondary symptom scored 0, 1, 2, 3 respectively according to severity of each symptom. Total symptom score represented the syndrome score. Change of the syndrome score from baseline was compared between treatment group and control group at different time windows. Reduction in syndrome score represented Improvement
Change of gastroesophageal Reflux Disease-Health Related Quality of Life (GERD-HRQL) scale score | week 2, week 4 during treatment period, week 6 and week 8 during follow-up period
  Gastroesophageal Reflux Disease-Health Related Quality of Life (GERD-HRQL) scale was used to evaluate the quality of life of patients with non-erosive reflux disease. Change of GERD-HRQL scale total score (0-55) from baseline was compared between treatment group and control group at different time windows. Reduction in total score represented Improvement
Change of patient ported outcome (PRO) for chronic gastrointestinal disease scale score | week 2, week 4 during treatment period, week 6 and week 8 during follow-up period
  Patient ported outcome (PRO) for chronic gastrointestinal disease scale was used to evaluate the efficacy of experimental drug. Change of PRO scale total score (0-152) from baseline was compared between treatment group and control group at different time windows. Reduction in total score represented Improvement
Change of self-rating anxiety scale (SAS) score | week 2, week 4 during treatment period, week 6 and week 8 during follow-up period
  Self-rating anxiety scale (SAS) was used to evaluate the efficacy of experimental drug. Change of SAS total score (20-80) from baseline was compared between treatment group and control group at different time windows. Reduction in total score represented Improvement
Change of self-rating depression scale (SDS) score | week 2, week 4 during treatment period, week 6 and week 8 during follow-up period
  Self-rating depression scale (SDS) was used to evaluate the efficacy of experimental drug. Change of SAS total score (20-80) from baseline was compared between treatment group and control group at different time windows. Reduction in total score represented Improvement

CONTACTS AND LOCATIONS:
Overall Officials: beihua zhang, M.D, Study Chair — Xiyuan Hospital of China Academy of Chinese Medical Sciences; guang bai, M.D, Study Director — Liaoning University of Traditional Chinese Medicine; wei wang, M.M, Study Director — First Teaching Hospital of Tianjin University of Traditional Chinese Medicine
Locations (1):
- Xiyuan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang T, Bai G, Wang W, Liu L, Zhou Z, Ji H, Zhang B, Tang X. Efficacy and safety of Jianpi Qinghua granules for non-erosive reflux disease with spleen deficiency and damp-heat syndrome: a multicenter, randomized, double-blind, placebo-controlled clinical trial. Front Nutr. 2025 Jan 7;11:1509931. doi: 10.3389/fnut.2024.1509931. eCollection 2024. PMID 39839278